CLINICAL TRIAL: NCT02645773
Title: Early Intervention With Non-ablative Fractional Laser to Reduce Cutaneous Scarring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Katrine Elisabeth Karmisholt, MD, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Early intevention
Record Dates: First submitted 2015-12-30; First posted 2016-01-05 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Cicatrix
MeSH Terms: conditions — Cicatrix | interventions — Lasers

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Pre-laser (Experimental): non-ablative laser Laser Pre-wounding low dose laser Pre-wounding medium dose laser Pre-wounding high dose
  Interventions: Device: non-ablative laser
- Immediate-laser (Experimental): non-ablative laser Laser low dose - immediate after wounding Laser medium dose - immediate after wounding Laser high dose - immediate after wounding
  Interventions: Device: non-ablative laser
- Post-laser (Experimental): non-ablative laser Laser low dose - post wounding Laser medium dose - post wounding Laser medium dose - post wounding
  Interventions: Device: non-ablative laser
- Control (No Intervention): Untreated control wound

INTERVENTIONS:
Device: non-ablative laser — non-abaltive laser pre, immediate and post wounding
  Other Names: Erbium:glass laser; 1540 nm laser
  Arms: Immediate-laser; Post-laser; Pre-laser

SUMMARY:
To investigate intervention with early application of non-ablative laser to prevent scarring in the skin

DETAILED DESCRIPTION:
To intervene in scar formation at three different time-points

ELIGIBILITY:
Inclusion Criteria:

* good health
* men
* Skin type 2-3
* non-smokers
* presenting full medical record

Exclusion Criteria:

* active skin disease in test area
* resent UV-exposure in test area
* history of keloid
* current or resent cancer
* uncontrolled systemical disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-09; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
To measure the clinical effect on scarring of non-ablative laser intervention at the three time-points | 3 months after
  Clinical evaluation by scar scales

CONTACTS AND LOCATIONS:
Overall Officials: Merete Haedersdal, professor, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark